CLINICAL TRIAL: NCT05452837
Title: Free Dermal Fat Graft (FDFG) Versus Superficial Musculoaponeurotic System (SMAS) Flap After Superficial Parotidectomy; Evaluation of Functional and Esthetic Outcome
Brief Title: FDFG Versus SMAS Flap After Superficial Parotidectomy; Evaluation of Functional and Esthetic Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, M. Ashraf Balbaa, Professor of Surgery, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7/2022SURG3B
Record Dates: First submitted 2022-06-16; First posted 2022-07-11 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Frey Syndrome
Keywords: Frey's syndrome; Postparotidectomy reconstruction
MeSH Terms: conditions — Sweating, Gustatory

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Dermal Fat Graft (Active Comparator): Free Dermal Fat Graft (FDFG) is applied to the superficial parotidectomy defect site
  Interventions: Procedure: FDFG
- Superficial musculoaponeurotic system flap (Active Comparator): Superficial musculoaponeurotic system (SMAS) Flap is dissected and tailored to fill the defect after superficial parotidectomy
  Interventions: Procedure: SMAS

INTERVENTIONS:
Procedure: FDFG — FDFG is applied to the parotidectomy bed after superficial parotidectomy
  Arms: Free Dermal Fat Graft
Procedure: SMAS — SMAS flap is applied to the parotidectomy bed after superficial parotidectomy
  Arms: Superficial musculoaponeurotic system flap

SUMMARY:
After parotidectomy, Frey's syndrome and facial disfigurement are the most common encountered complications. Free dermal fat graft (FDFG) and the superficial musculoaponeurotic system (SMAS) flap, have very promising results. In this study, the functional and esthetic outcome from their usage were compared.

DETAILED DESCRIPTION:
Parotidectomy is the standard procedure for treatment of many parotid lesions, however it carries a lot of drawbacks. Facial asymmetry and Frey's syndrome are the most annoying complications to the patients. Insertion of inter-positioning grafts at parotidectomy bed can decrease these complications significantly. Free dermal fat graft (FDFG) and the superficial musculoaponeurotic system (SMAS) flap, have very promising results. In this study the investigators have compared the functional and esthetic outcome from their usage.

Seventy-eight patient underwent parotidectomy for various causes. The patients were divided randomly in 2 groups each group 39 patients. In one group FDFG was inserted at the parotidectomy bed, while in the other group SMAS flap was performed. Preoperative, operative, and postoperative data were recorded and analyzed.

The normality of distribution of variables was verified by Wilks -Shapiro test. The data were expressed as Number (No), percentage (%) mean (x̅) and standard deviation (SD). Chi-square test (χ2) was used to study association between qualitative variables. Whenever any of the expected cells were less than five, Fischer's Exact test was used. Student's t-test is a test of significance used for comparison of quantitative variables between two groups of normally distributed data, while Mann Whitney's test was used for comparison of quantitative variables between two groups of not normally distributed data. Two-sided P value was set to be significant if < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for superficial parotidectomy

Exclusion Criteria:

* Less than 18 years of age
* Proved malignant parotid tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with Frey's syndrome | 6 months
  Number of patients who developed of Frey's syndrome as post-parotidectomy complication

SECONDARY OUTCOMES:
Degree of patients' satisfaction with the fascial symmetry | 6 months
  Assessment of degree of patients' satisfaction of the esthetic outcome after parotidectomy regarding post parotidectomy facial symmetry based on a verbal descriptive scale; excellent, good, fair, and poor. It is not based on numerical scale.
  Number of patients who will have excellent, good, fair or poor response will be recorded and compared within the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: M. Ashraf Balbaa, M.D., Principal Investigator — Faculty of Medicine, Menoufia University
Locations (1):
- Faculty of Medicine, Menoufia University, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be available to be shared on request after study publication for 6 months.
Supporting Information: Study Protocol, SAP
Time Frame: Six months from the time of study publication
Access Criteria: Contacting the corresponding author

REFERENCES:
- [Result] Curry JM, King N, Reiter D, Fisher K, Heffelfinger RN, Pribitkin EA. Meta-analysis of surgical techniques for preventing parotidectomy sequelae. Arch Facial Plast Surg. 2009 Sep-Oct;11(5):327-31. doi: 10.1001/archfacial.2009.62. PMID 19797095
- [Derived] Fawzy A, Balbaa MA, Hagag M. Evaluation of functional and aesthetic outcomes of free dermal fat graft versus superficial musculoaponeurotic system flap after superficial parotidectomy: randomized clinical trial. BJS Open. 2023 May 5;7(3):zrac173. doi: 10.1093/bjsopen/zrac173. PMID 37151084